CLINICAL TRIAL: NCT04985851
Title: Durvalumab (MEDI4736) Combined With Anlotinib Versus Durvalumab (MEDI4736) Alone as Maintenance Therapy in Extensive-Stage Small-Cell Lung Cancer (ES-SCLC)
Brief Title: To Evaluate the Efficacy of Durvalumab + Anlotinib in Terms of OS and PFS.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, Chief physician, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-20-20841
Record Dates: First submitted 2021-06-07; First posted 2021-08-02 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Extensive-Stage Small-Cell Lung Cancer
Keywords: Durvalumab; Extensive-Stage Small-Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab; anlotinib

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomised, multicenter, Phase II study. This study is planned to enroll 90 eligible patients to receive durvalumab combined with up to 4 cycles of etoposide and platinum-based chemotherapy (EP). And approximately 64 patients who complete the 4 cycles of durvalumab + EP treatment and don't have progressive diseases (Non-PD patients) will be randomized in a 1:1 ratio to receive maintenance treatment durvalumab + anlotinib (Arm 1) or durvalumab (Arm 2) until confirmed progressive disease. Prophylactic cranial irradiation (PCI) is allowed at the investigators' discretion as per SoC guidance for ES-SCLC. Patients will attend a safety follow up visit 90 days after last dose of durvalumab
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- maintenance treatment durvalumab + anlotinib (Experimental): Durvalumab 1500 mg monotherapy will be continued q4w. Anlotinib will be administered according to prescribing information in general use. The dose is 12mg, QD, PO, 14 days-on and 7 days-off.
  * N.B. If a patient's weight falls to 30 kg or below (≤30 kg) the patient should receive weight-based dosing equivalent to 20 mg/kg of durvalumab until the weight improves to >30 kg, at which point the patient should start receiving the fixed dosing of durvalumab 1500 mg.
  * Anlotinib is available at three dose levels, 12 mg, 10 mg, and 8 mg. Dose reduction may take place whenever toxicity that is not controlled with optimal supportive care is noted during the study. If a subject subsequently tolerates treatment well at that level in the judgment of the investigator, the dose may be increased to the next dose level. If a subject cannot tolerate treatment after dose reduction to 8 mg, treatment will be discontinued
  Interventions: Drug: durvalumab + anlotinib
- maintenance treatment durvalumab (Active Comparator): Durvalumab 1500 mg monotherapy will be continued q4w.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: durvalumab + anlotinib — Approximately 64 patients who complete the 4 cycles of durvalumab + EP treatment and don't have progressive diseases (Non-PD patients) will be randomized in a 1:1 ratio to receive maintenance treatment durvalumab + anlotinib (Arm 1) or durvalumab (Arm 2) until confirmed progressive disease.
  Arms: maintenance treatment durvalumab + anlotinib
Drug: Durvalumab — durvalumab
  Arms: maintenance treatment durvalumab

SUMMARY:
This is an open-label, randomised, multicenter, Phase II study. This study is planned to enroll 90 eligible patients to receive durvalumab combined with up to 4 cycles of etoposide and platinum-based chemotherapy (EP). And approximately 64 patients who complete the 4 cycles of durvalumab + EP treatment and don't have progressive diseases (Non-PD patients) will be randomized in a 1:1 ratio to receive maintenance treatment durvalumab + anlotinib (Arm 1) or durvalumab (Arm 2) until confirmed progressive disease. Prophylactic cranial irradiation (PCI) is allowed at the investigators' discretion as per SoC guidance for ES-SCLC. Patients will attend a safety follow up visit 90 days after last dose of durvalumab. Tumor assessments will be performed at Screening with follow-up at Week 6 ±1 week and Week 12 ±1 week from the date of the first cycle treatment, and then every 8 weeks ±1 week until confirmed objective disease progression.

DETAILED DESCRIPTION:
Target subject population Adult patients (aged ≥18 years) with histologically or cytologically documented extensive disease (American Joint Committee on Cancer Stage (8th edition) IV SCLC [T any, N any, M1 a/b]), or T3-4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan. Patients must have World Health Organization/Eastern Cooperative Oncology Group performance status of 0-1, weight > 30 kg and adequate organ and marrow function. All patients are suitable for firstline platinum-based chemotherapy.

Duration of treatment Unless specific treatment discontinuation criteria are met, patients in Arms 1 and 2 will continue therapy until disease progression, as per investigator assessment. Investigational product, dosage and mode of administration Durvalumab 1500 mg will be administered for all patients via IV infusion concurrently with EP q3w starting on week 0 for 4 cycles. Non-PD patients who completed the 4 cycles of Durvalumab + EP will be randomized 1:1 into Arm 1 and Arm 2. Eligible patients should begin continuous treatment in 3 days after randomization.

* Arm 1: Durvalumab 1500 mg monotherapy will be continued q4w. Anlotinib will be administered according to prescribing information in general use. The dose is 12mg, QD, PO, 14 days-on and 7 days-off.
* N.B. If a patient's weight falls to 30 kg or below (≤30 kg) the patient should receive weight-based dosing equivalent to 20 mg/kg of durvalumab until the weight improves to >30 kg, at which point the patient should start receiving the fixed dosing of durvalumab 1500 mg. Anlotinib is available at three dose levels, 12 mg, 10 mg, and 8 mg. Dose reduction may take place whenever toxicity that is not controlled with optimal supportive care is noted during the study. If a subject subsequently tolerates treatment well at that level in the judgment of the investigator, the dose may be increased to the next dose level. If a subject cannot tolerate treatment after dose reduction to 8 mg, treatment will be discontinued.
* Arm 2: Durvalumab 1500 mg monotherapy will be continued q4w.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤75 years
* Histologically or cytologically documented extensive disease (American Joint Committee on Cancer Stage (8th edition) IV SCLC [T any, N any, M1 a/b/c]), or T3-4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan.
* Brain metastases must be asymptomatic or treated and stable off steroids and anti convulsants for at least 1 month prior to study treatment. Patients with suspected brain metastases at screening should have a CT/MRI of the brain prior to study entry.
* Having at least one measurable lesion according to RECIST 1.1.
* No prior systemic therapy for ES-SCLC
* Suitable to receive a platinum (cisplatin or carboplatin) based chemotherapy regimen as 1st-line treatment for the ES-SCLC.
* ECOG PS score: 0 to 1
* Life expectancy ≥ 12 weeks.
* Body weight > 30kg
* No prior exposure to immune-mediated therapy including, but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines.
* No prior exposure to anti-angiogenesis drugs.
* Adequate organ and marrow function as defined below:

Absolute neutrophil count ≥1.5×109 /L, platelet count≥100 ×109 /L, hemoglobin ≥9.0g/dL [no blood transfusion or no erythropoietin (EPO) dependence within 7 days before enrollment]. Biochemical test results should meet the following criteria: Serum bilirubin < 1.5 times the upper limit of normal value (ULN); ALT and AST < 2.5 × ULN; in case of liver metastases, ALT and AST < 5 × ULN; Creatinine clearance (CCr) >60ml/min for patients on cisplatin and >45ml/min for patients on carboplatin, as determined by Cockcroft-Gault (using actual body weight);

* International normalized ratio (INR) and prothrombin time (PT) ≤1.5 times ULN for patients not receiving therapeutic anticoagulation
* Women of child-bearing age should agree to take contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study and within 6 months after the study; non-breast-feeding patients whose serum or urinary pregnancy test should be negative; male patients should agree to take contraceptive measures during the study and within 6 months after the study.
* Patients are voluntarily enrolled into the study, sign the informed consent form and have good compliance.

Exclusion Criteria:

* Previous IP assignment in the present study;
* Concurrent enrolment in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study.
* Patients with inability to take oral medication, including but not limited to dysphagia, gastrointestinal resection, chronic diarrhea and intestinal obstruction;
* Any history of radiotherapy to the chest prior to systemic therapy or planned consolidation chest radiation therapy. Radiation therapy outside of the chest for palliative care (ie, bone metastasis) is allowed but must be completed before first dose of the study medication.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogeneic organ transplantation.
* Has a paraneoplastic syndrome (PNS) of autoimmune nature, requiring systemic treatment (systemic steroids or immunosuppressive agents) or has a clinical symptomatology suggesting worsening of PNS.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis with the exception of diverticulosis, systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, and uveitis, etc]). The following are exceptions to this criterion: Patients with vitiligo or alopecia; Patients with hypothyroidism (eg, following Hashimoto syndrome) and stable on hormone replacement; Any chronic skin condition that does not require systemic therapy; Patients without active disease in the last 5 years may be included but only after consultation with the Study Physician; Patients with celiac disease controlled by diet alone
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive HBV surface antigen [HbsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HbsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion: Intranasal, inhaled, topical steroids or local steroid injections (eg, intra articular injection); Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent; Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication). Premedication with steroids for chemotherapy is acceptable.
* History of active primary immunodeficiency.
* Patients who are known to have symptomatic brain metastases or carcinomatous meningitis, or brain or leptomeningeal disease diagnosed by CT or MRI at the time of screening;
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of IP. Note:

Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.

* Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses (<30 mm from the carina) of large volume.
* Evidence of bleeding diathesis or significant coagulopathy (in absence of therapeutic anticoagulation)
* Not completely controlled eye inflammation or eye infection, or any condition that may lead to the above-mentioned ocular diseases
* Patients with any severe and/or unable to control diseases，including： Interstitial lung disease Blood pressure unable to be controlled ideally(systolic pressure>140 mmHg， diastolic pressure>90 mmHg); Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QTc≥450ms(male),QTc≥470ms（female）) and patients with Grade 1 or higher congestive heart failure (NYHA Classification); Patients with cirrhosis, decompensated liver disease, or active hepatitis; Patients with poorly controlled diabetes (fasting blood glucose(FBG)>10mmol/L) Serious chronic gastrointestinal conditions associated with diarrhea Urine protein ≥ ++，and 24-hour urinary protein excretion>1.0 g confirmed; Psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* Uncontrolled hypercalcemia (> 1.5 mmol/L calcium ion or calcium > 12 mg/dL or corrected serum calcium > ULN), or symptomatic hypercalcemia requiring continued diphosphate therapy;
* Patients with unhealed wounds or fractures;
* Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism
* Patients who are known to have severe allergies (≥ grade 3) to active ingredients and any excipients of anlotinib or durvalumab;
* Patients who have other malignant tumors (except radical cervical carcinoma in situ, non-melanoma skin cancer, etc.) at the same time;
* The subjects or their sexual partners cannot or refuse to take effective contraceptive measures during the clinical trial
* Pregnant or breast-feeding womenPatients in other situations who are evaluated by the investigator to be ineligible to be enrolled.Procedures for withdrawal of incorrectly enrolled subjects see Section 3.4

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS-Progression Free Survival | 2 years
  The time from the start of systemic treatment date to the date of first documented disease progression (event: disease progression - DP, based on RECIST, death, adverse events, which provide to disqualification from further therapy).

SECONDARY OUTCOMES:
OS-Overall Survival | 2 years
  The time from the start of systemic treatment date to the date of death due to any cause or the date of last contact (censored observation) at the date of data cut-off

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China